CLINICAL TRIAL: NCT06481787
Title: A Single-centre Randomised Controlled Study of 8-week Zuojinwan in Combination With Volnoxan Fumarate for the Treatment of Gastro-oesophageal Reflux Disease Combined With Depression
Brief Title: Zuojin Wan Combined With Woonosan Fumarate for the Treatment of GRD Combined With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KY20240613-03-KS-01
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Gastroesophageal Reflux Disease; Depression
MeSH Terms: conditions — Gastroesophageal Reflux; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonorasan fumarate (Experimental): Vonorasan fumarate, 20 mg twice daily orally before meals for 8 weeks of treatment.
  Interventions: Drug: Vonorasan Fumarate
- Zuojin Pills combined with Vonorasan Fumarate (Experimental): Add Zuojin Pills, 3g each time, twice daily, on top of Vonorasan Fumarate treatment for 8 weeks.
  Interventions: Drug: Vonorasan Fumarate; Drug: Zuojin Pills

INTERVENTIONS:
Drug: Vonorasan Fumarate — Vonorasan fumarate is taken 30min before breakfast and dinner.
Drug: Zuojin Pills — Zuojin Pills should be taken 30min after breakfast and dinner.
  Arms: Zuojin Pills combined with Vonorasan Fumarate

SUMMARY:
To evaluate the improvement of symptoms in patients with gastroesophageal reflux disease combined with depression (hepatic and gastric depression-heat type) by Zuojin Wan combined with vornodine fumarate regimen as a control, and to compare the adherence to the medication and the adverse reactions of the patients between the two groups.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a common digestive disorder, and in recent years studies have shown an increasing incidence of comorbid depression in patients with GERD. The treatment of gastric acid inhibition and mucosal protection alone is not effective for patients with reflux combined with depression, and the additional administration of neuromodulatory drugs will increase the incidence of adverse reactions, so the combination of traditional Chinese medicine may be one of the effective ways to solve the above problems. The aim of this study was to compare the efficacy of Zuojin Wan combined with vunorasan fumarate with that of vunorasan fumarate alone.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years;
2. Fulfilment of western medical diagnostic criteria for GERD;
3. Meet the diagnostic criteria for mild depression;
4. Comply with the diagnostic criteria of Liver and Stomach Depression-Heat syndrome in Chinese medicine;
5. A score of 7-17 on the 17-item Hamilton Depression Scale (HAMD-17) (7-17 being mild depression);
6. Good compliance and autonomous behaviour;
7. No medications that may have an effect on the study, such as acid-suppressing agonists, were taken within 2 weeks prior to enrolment;

Exclusion Criteria:

1. HP positive patients;
2. Other organic diseases of the digestive system, such as peptic ulcer, peptic tumour, peptic haemorrhage, liver, gallbladder and pancreas disease, intestinal obstruction and inflammatory bowel disease;
3. Systemic diseases affecting the dynamics of the digestive tract, such as diabetes mellitus, chronic renal insufficiency, connective tissue diseases, neurological lesions, etc;
4. Pathological diagnosis of the esophageal mucosa suggestive of moderate-to-severe heterogeneous hyperplasia;
5. Previous surgery resulting in a decrease in gastric acid or a history of oesophageal or gastric surgery;
6. Varicose veins in the esophagus or fundus of the stomach;
7. Persons with severe primary heart, brain, liver, lung, kidney, blood or serious disease affecting their survival;
8. Those with depression, suicidal tendencies and mental disorders who cannot cooperate;
9. Pregnant or breastfeeding women, or patients who have a plan to have children in the near future;
10. Taking drugs that have an effect on the results of this study within 2 weeks before participating in this study;
11. Allergy or adverse reaction to the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reflux Disease Questionnaire | Baseline and 8 weeks
  According to the frequency and severity of episodes of the main symptoms，observe the changes of reflux'disease questionnaire score before treatment and after 8 weeks of treatment.
Hamilton Depression Scale | Baseline and 8 weeks
  Assessing patients for depressive symptoms
Chinese Medicine Points Scale | Baseline and 8 weeks
  Assessment of TCM evidence before and after treatment

SECONDARY OUTCOMES:
Adverse events during treatment | Baseline and 8 weeks
  Ask the patient about the occurrence of adverse events while taking the medication

CONTACTS AND LOCATIONS:
Overall Officials: wanli liu, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No